CLINICAL TRIAL: NCT07010237
Title: Dose-attenuated IST and Hetrombopag in the Treatment of Elderly (≥65 Years) Patients With Very Severe/Severe Aplastic Anemia: A Single-Center, Single-Arm, Phase IIB Clinical Study on Efficacy and Safety
Brief Title: Dose-attenuated IST and Hetrombopag in Elderly (≥65 Years) Patients With Severe Aplastic Anemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025013
Record Dates: First submitted 2025-04-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-02

CONDITIONS: Sever Aplastic Anaemia; Elderly (People Aged 65 or More); Immunosuppressive Treatment
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A-IST (Experimental): Porcine-ATG : 15 mg/kg/day IV ×5 days. Cyclosporine : 3-5 mg/kg/day (adjusted to trough 100-200 μg/L). Hetrombopag: 15 mg daily.
  Interventions: Drug: Dose-attenuated IST and Hetrombopag

INTERVENTIONS:
Drug: Dose-attenuated IST and Hetrombopag — Porcine-ATG : 15 mg/kg/day IV ×5 days. Cyclosporine : 3-5 mg/kg/day (adjusted to trough 100-200 μg/L). Hetrombopag: 15 mg daily for 24weeks.

SUMMARY:
This is a prospetive,Single-Center, Single-Arm, Phase IIB Clinical Study.This study aims to evaluate the efficacy and safety of dose-attenuated IST combined with Hetrombopag in elderly patients (≥65 years) with VSAA/SAA.

DETAILED DESCRIPTION:
Design : Prospective, single-center, single-arm, open-label Phase IIB trial.

Intervention :

P-ATG : 15 mg/kg/day IV ×5 days. Cyclosporine : 3 mg/kg/day (adjusted to trough 100-200 μg/L). Hetrombopag : 15 mg daily. Follow-Up : Weekly for 24 weeks, with bone marrow evaluation at 24 weeks.

Inclusion Criteria :

Confirmed diagnosis of VSAA/SAA. Age ≥65 years. Completion of all screening assessments. Ability to swallow oral medication. Signed informed consent (by patient or legal guardian if patient is incapacitated).

Exclusion Criteria :

Clonal cytogenetic abnormalities (excluding isolated -Y or +8). Prior treatment with ATG/high-dose cyclophosphamide. Prior cyclosporine/tacrolimus use >12 months. Prior TPO-RA therapy >3 months. Uncontrolled malignancies or conditions contraindicating ATG. Severe organ dysfunction (e.g., creatinine ≥177 μmol/L). Investigator judgment of unsuitability.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of VSAA/SAA.
* Age ≥65 years.
* Completion of all screening assessments.
* Must be able to swallow tablets.
* Signed informed consent (by patient or legal guardian if patient is incapacitated).

Exclusion Criteria:

* Clonal cytogenetic abnormalities (excluding isolated -Y or +8).
* Prior treatment with ATG/high-dose cyclophosphamide.
* Prior cyclosporine/tacrolimus use >12 months.
* Prior TPO-RA therapy >3 months.
* Uncontrolled malignancies or conditions contraindicating ATG.
* Severe organ dysfunction (e.g., creatinine ≥177 μmol/L).
* Investigator judgment of unsuitability.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Hematologic response rate at 24 weeks post-ATG treatment. | 24 weeks
  PR+CR Partial Response (PR) : Independence from transfusions without meeting CR. No Response (NR) : Failure to achieve PR.

SECONDARY OUTCOMES:
Early mortality rate | 12 weeks
  Early mortality rate within 12weeks
Complete Response | 24 weeks
  Complete Response (CR) : HGB ≥100 g/L, PLT ≥100×10⁹/L, ANC ≥1.0×10⁹/L.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, CAMS
Locations (1):
- Red Blood Cell Diseases Center, Tianjin, Tianjin Municipality, China